CLINICAL TRIAL: NCT05066230
Title: A Prospective, Randomized, Double-masked, Sham-controlled, Multicenter, Two-arm Phase3 Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 in Participants With Moderately Severe to Severe Non-proliferative Diabetic Retinopathy
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravitreal KSI-301 in Non-proliferative Diabetic Retinopathy (NPDR)
Acronym: GLOW
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: All patients completed the primary endpoint assessments. Additional follow-up after the primary endpoint was deemed not necessary by the Sponsor.
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS301P106
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Non-proliferative Diabetic Retinopathy
Keywords: Non-proliferative Diabetic Retinopathy; Diabetic Retinopathy; NPDR; KSI-301; VEGF; Anti-VEGF; Vascular Endothelial Growth Factor; Antibody Biopolymer Conjugate; Retinal Degeneration; Retinal Diseases; Eye Diseases; Retinopathy; Vision Disorders; Kodiak
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Degeneration; Retinal Diseases; Eye Diseases; Vision Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two arms: KSI-301 or sham.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: To preserve masking, 2 investigators are required for this study. The masked investigator will be responsible for examinations and safety assessments. The unmasked investigator will perform the injections and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 - Treatment Group A (Experimental): Intravitreal injection of KSI-301 (5 mg): three initiating doses, and then every 24 weeks through Week 92
  Interventions: Drug: KSI-301
- Treatment Group B (Sham Comparator): Sham injection on the same schedule as Treatment Group A
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: KSI-301 — Intravitreal injection
  Arms: KSI-301 - Treatment Group A
Other: Sham injection — The sham injection is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It is performed to maintain masking of the study.
  Arms: Treatment Group B

SUMMARY:
This Phase 3 Study will evaluate the efficacy and safety of KSI-301 in participants with moderately severe to severe non-proliferative diabetic retinopathy (NPDR).

DETAILED DESCRIPTION:
This is a Phase 3, prospective, randomized, double-masked, sham-controlled, two-arm, multicenter study evaluating the efficacy and safety of repeated intravitreal dosing of KSI-301 5 mg in participants with moderately severe to severe non-proliferative diabetic retinopathy (NPDR).

The primary endpoint will be assessed at Week 48; additional secondary endpoints for efficacy will be assessed at Week 48, Week 96 and if applicable, over time.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to participation in the study.
* Type 1 or 2 diabetes mellitus
* Moderately severe to severe NPDR in the Study Eye (DRSS levels 47 and 53 as determined by the reading center), in which pan-retinal photocoagulation (PRP) can be safely deferred for at least 6 months per the Investigator.
* BCVA ETDRS letter score in the Study Eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better)
* HbA1c of ≤12%.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Presence of center-involved DME in the Study Eye
* Prior PRP in the Study Eye.
* Current anterior segment neovascularization (ASNV), vitreous hemorrhage, or tractional retinal detachment in the Study Eye.
* Prior intravitreal anti-VEGF treatment in the Study Eye for DR or DME.
* Prior intravitreal or periocular steroid in the Study Eye for DR or DME.
* Prior use of an investigational intravitreal treatment for DR or DME in the Study Eye.
* Any history or evidence of a concurrent ocular condition present in the Study Eye, that in the opinion of the Investigator could require either medical or surgical intervention or alter visual acuity during the study
* Active or suspected ocular or periocular infection or inflammation.
* Women who are pregnant or lactating or intending to become pregnant during the study.
* History of a medical condition that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product.
* Recent history (within the 6 months prior to screening) of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure or any acute coronary event.
* Uncontrolled blood pressure defined as a systolic value ≥ 180 mmHg or diastolic value ≥ 100 mmHg while at rest.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc; Daniel Janer, MD, Study Director — Kodiak Sciences Inc
Locations (61):
- United States (46):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Vitreous Associates, Beverly Hills, California
  - Retina Consultants of Orange County, Fullerton, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Connecticut Eye Consultants, Danbury, Connecticut
  - Retina Group of New England, Waterford, Connecticut
  - The Macula Center/ Blue Ocean Clinical Research, Clearwater, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Med Eye Associates, Miami, Florida
  - Florida Retina Institute, Orlando, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Retina Specialists of Idaho, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Retina Associates PA, Lenexa, Kansas
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular LLC, Bloomfield, New Jersey
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Graystone Eye, Hickory, North Carolina
  - Cascade Medical Research Institute, Eugene, Oregon
  - MidAtlantic Retina, Bethlehem, Pennsylvania
  - Charleston Neurosciences Institute, Beaufort, South Carolina
  - Charleston Neuroscience Center, Charleston, South Carolina
  - Southeastern Retina Associates PC, Knoxville, Tennessee
  - Charles Retina Institute, Memphis, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Panhandle Eye Group, LLP, Amarillo, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas (Houston), Bellaire, Texas
  - Star Vision Consultants, Burleson, Texas
  - Retina Consultants of Texas (Katy), Katy, Texas
  - Texas Retina Associates, Plano, Texas
  - Austin Retina Associates (Round Rock), Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Texas - (Woodlands), The Woodlands, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Spokane Eye, Spokane, Washington
- Czechia (2):
  - OFTEX s.r.o., Pardubice, Pardubický kraj
  - Axon Clinical, s.r.o., Prague
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Latvian American Eye Center, Riga
- Poland (3):
  - Warszawski Szpital Okulistyczny, Warsaw, Masovian Voivodeship
  - Optimum Profesorskie Centrum Okulistyki, Gdansk, Pomeranian Voivodeship
  - Oftalmika Sp. z o.o., Bydgoszcz
- Emanuelli Research & Development Center LLC, Arecibo, Puerto Rico
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F. D. Roosevelta, Banská Bystrica
  - Fakultna nemocnica Trencin, Trenčín
- Spain (5):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari General de Catalunya - Grupo Quironsalud, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid, Majadanonda
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 52 medical centers between September 2021 and August 2022. The first participant was enrolled on 07 September 2021 and the last on 25 August 2022.
Pre-assignment Details: Of 560 screened participants, 253 met eligibility criteria and were randomized to treatment.
Period: Primary Study (Through Week 48)
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Started | 128 | 125
Completed (Completed is defined as those who completed study through Week 48.) | 120 | 115
Not Completed | 8 | 10
Not completed — Adverse Event | 1 | 4
Not completed — Non-compliance with study schedule | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 2 | 3
Not completed — Participant relocated | 1 | 0
Period: After Week 48
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Started | 120 | 115
Completed (The study was discontinued by the Sponsor after all patients completed the primary endpoint assessment at Week 48.) | 0 | 0
Not Completed | 120 | 115
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with study schedule | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Sponsor Request | 115 | 111

BASELINE CHARACTERISTICS:
Population: Full analysis set defined as all randomized subjects who received any study treatment (KSI-301 or sham) and have gradable DRSS value at baseline. Subjects will be analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B | Total
Number analyzed (Participants) | 128 | 125 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 95 | 191
  >=65 years | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (11.39) | 57 (9.63) | 56.7 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 56 | 107
  Male | 77 | 69 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 52 | 109
  Not Hispanic or Latino | 71 | 73 | 144
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 23 | 36
  White | 108 | 96 | 204
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 3
Geographic Region [Count of Participants; unit: Participants]
  North America | 123 | 120 | 243
  Rest of World | 5 | 5 | 10
Diabetic Retinopathy Severity Scale (DRSS) at Baseline [Count of Participants; unit: Participants] — The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
  Participants
    DRSS Level ≤47 | 46 | 45 | 91
    DRSS Level ≥53 | 82 | 80 | 162

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Improving ≥2 Steps on DRSS
Description: Percentage of patients improving ≥2 steps on the Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 48 using last observation carried forward (LOCF). The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 52 | 2
Statistical Analysis 1: Comparison: KSI-301 - Treatment Group A vs Treatment Group B; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haentzel test stratified by baseline DRSS level (≤level 47 vs. ≥level 53) and HbA1c level (≤8.5% vs. >8.5%); Difference of weighted percentages = 39.7, 95.02% CI 2-sided [31.3 to 48.1] — Weighted percentages are based on weighted average of observed estimates across strata using CMH weights. The CI are based on the normal approximation to the binomial proportions

2. Secondary Outcome: Percentage of Patients Developing Any Sight-Threatening Complication
Description: Percentage of patients developing any of the following Sight-Threatening Complication: Proliferative Diabetic Retinopathy (PDR), Anterior segment neovascularization (ASNV), Vitreous hemorrhage or tractional retinal detachment believed to be due to PDR, or Diabetic Macular Edema (DME) from baseline through Week 48
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 3 | 26
Statistical Analysis 1: Comparison: KSI-301 - Treatment Group A vs Treatment Group B; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference of weighted percentages = -18.7, 95.02% CI 2-sided [-26.2 to -11.2] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Patients Improving ≥3 Steps on DRSS
Description: Percentage of patients improving ≥3 steps on the Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 48 using last observation carried forward (LOCF). The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 7 | 0
Statistical Analysis 1: Comparison: KSI-301 - Treatment Group A vs Treatment Group B; Test type: Superiority; p = 0.0058, Cochran-Mantel-Haenszel; Cochran-Mantel-Haentzel test stratified by baseline DRSS level (≤level 47 vs. ≥level 53), HbA1c level (≤8.5% vs. >8.5%); Difference of weighted percentages = 5.6, 95.02% CI 2-sided [1.6 to 9.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Patients Developing PDR
Description: Percentage of patients developing Proliferative Diabetic Retinopathy (PDR) from baseline through Week 48
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 2 | 10
Statistical Analysis 1: Comparison: KSI-301 - Treatment Group A vs Treatment Group B; Test type: Superiority; p = 0.0149, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference of weighted percentages = -6.5, 95.02% CI 2-sided [-11.8 to -1.3] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Patients Developing PDR or ASNV
Description: Percentage of patients developing Proliferative Diabetic Retinopathy (PDR) or Anterior segment neovascularization (ASNV) from baseline through Week 48
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 2 | 10

6. Secondary Outcome: Percentage of Patients Developing Vitreous Hemorrhage or Tractional Retinal Detachment Believed to be Due to PDR
Description: Percentage of patients developing vitreous hemorrhage or tractional retinal detachment believed to be due to Proliferative Diabetic Retinopathy (PDR) from baseline through Week 48
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 2 | 3

7. Secondary Outcome: Percentage of Patients Developing DME
Description: Percentage of patients developing Diabetic Macular Edema (DME) from baseline through Week 48
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants | 1 | 17

8. Secondary Outcome: Percentage of Patients With a ≥2-step or ≥3-step Worsening on DRSS
Description: Percentage of patients with a ≥2-step or ≥3-step worsening on the Diabetic Retinopathy Severity Scale (DRSS) from baseline at Week 48 using last observation carried forward (LOCF). The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Severity range from level 10 (DR absent) to level 85 (advanced proliferative DR: posterior fundus obscured, or center of macula detached).
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants
  Patients with a ≥2-step worsening on DRSS | 1 | 5
  Patients with a ≥3-step worsening on DRSS | 0 | 3

9. Secondary Outcome: Percentage of Patients Who Lost ≥5, ≥10, or ≥15 Letters in BCVA
Description: Percentage of patients who lost ≥5, ≥10, or ≥15 letters in Best-corrected Visual Acuity (BCVA) from baseline by visit over time. Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Day 1 to Week 48
Population: Full analysis set defined as all randomized subjects who received any study treatment (KSI-301 or sham) and have gradable DRSS value at baseline. Subjects will be analyzed according to their randomized treatment. The Overall Number of Participants Analyzed were 128 and 125, but the number analyzed for each row is different depending on the number of participants with data for that row.
Measure: Count of Participants; unit: Participants
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Participants
  Participants who lost ≥ 5 letters from baseline to Week 8: number analyzed (Participants) | 127 | 123
  Participants who lost ≥ 5 letters from baseline to Week 8 | 8 | 15
  Participants who lost ≥ 5 letters from baseline to Week 20: number analyzed (Participants) | 122 | 109
  Participants who lost ≥ 5 letters from baseline to Week 20 | 15 | 15
  Participants who lost ≥ 5 letters from baseline to Week 32: number analyzed (Participants) | 117 | 99
  Participants who lost ≥ 5 letters from baseline to Week 32 | 17 | 10
  Participants who lost ≥ 5 letters from baseline to Week 44: number analyzed (Participants) | 109 | 90
  Participants who lost ≥ 5 letters from baseline to Week 44 | 12 | 8
  Participants who lost ≥ 5 letters from baseline to Week 48: number analyzed (Participants) | 114 | 91
  Participants who lost ≥ 5 letters from baseline to Week 48 | 14 | 11
  Participants who lost ≥ 10 letters from baseline to Week 8: number analyzed (Participants) | 127 | 123
  Participants who lost ≥ 10 letters from baseline to Week 8 | 2 | 3
  Participants who lost ≥ 10 letters from baseline to Week 20: number analyzed (Participants) | 122 | 109
  Participants who lost ≥ 10 letters from baseline to Week 20 | 2 | 4
  Participants who lost ≥ 10 letters from baseline to Week 32: number analyzed (Participants) | 117 | 99
  Participants who lost ≥ 10 letters from baseline to Week 32 | 5 | 1
  Participants who lost ≥ 10 letters from baseline to Week 44: number analyzed (Participants) | 109 | 90
  Participants who lost ≥ 10 letters from baseline to Week 44 | 4 | 2
  Participants who lost ≥ 10 letters from baseline to Week 48: number analyzed (Participants) | 114 | 91
  Participants who lost ≥ 10 letters from baseline to Week 48 | 5 | 1
  Participants who lost ≥ 15 letters from baseline to Week 8: number analyzed (Participants) | 127 | 123
  Participants who lost ≥ 15 letters from baseline to Week 8 | 1 | 1
  Participants who lost ≥ 15 letters from baseline to Week 20: number analyzed (Participants) | 122 | 109
  Participants who lost ≥ 15 letters from baseline to Week 20 | 1 | 1
  Participants who lost ≥ 15 letters from baseline to Week 32: number analyzed (Participants) | 117 | 99
  Participants who lost ≥ 15 letters from baseline to Week 32 | 4 | 0
  Participants who lost ≥ 15 letters from baseline to Week 44: number analyzed (Participants) | 109 | 90
  Participants who lost ≥ 15 letters from baseline to Week 44 | 0 | 0
  Participants who lost ≥ 15 letters from baseline to Week 48: number analyzed (Participants) | 114 | 91
  Participants who lost ≥ 15 letters from baseline to Week 48 | 3 | 0

10. Secondary Outcome: Time to First Development of PDR, ASNV, or DME
Description: Time to first development of Proliferative Diabetic Retinopathy (PDR), Anterior segment neovascularization (ASNV), or Diabetic Macular Edema (DME) through Week 48
Time Frame: Day 1 to Week 48
Population: Full analysis set defined as all randomized subjects who received any study treatment (KSI-301 or sham) and have gradable DRSS value at baseline. Subjects will be analyzed according to their randomized treatment. Subjects who did not have an event were censored at the date of the last scheduled study visit at or prior to Week 48.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Months | NA [NA to NA] — NA = Not available due to small number of PDR, ASNV, and DME events | NA [11.5 to NA] — NA = Not available due to small number of PDR, ASNV, and DME events

11. Secondary Outcome: Time to First Development of PDR or ASNV
Description: Time to first development of Proliferative Diabetic Retinopathy (PDR) or Anterior segment neovascularization (ASNV) through Week 48
Time Frame: Day 1 to Week 48
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Months | NA [NA to NA] — NA = Not available due to small number of PDR and ASNV events | NA [11.5 to NA] — NA = Not available due to small number of PDR and ASNV events

12. Secondary Outcome: Time to First Development of Vitreous Hemorrhage or Tractional Retinal Detachment Believed to be Due to PDR
Description: Time to first development of vitreous hemorrhage or tractional retinal detachment believed to be due to Proliferative Diabetic Retinopathy (PDR) through Week 48
Time Frame: Day 1 to Week 48
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Months | NA [NA to NA] — NA = Not available due to small number of vitreous hemorrhage and tractional retinal detachment events | NA [NA to NA] — NA = Not available due to small number of vitreous hemorrhage and tractional retinal detachment events

13. Other Pre Specified Outcome: Time to First Development of DME
Description: Time to first development of Diabetic Macular Edema (DME) through Week 48
Time Frame: Day 1 to Week 48
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Months | NA [NA to NA] — NA = Not available due to small number of DME events | NA [NA to NA] — NA = Not available due to small number of DME events

14. Other Pre Specified Outcome: Mean Change in OCT CST
Description: Mean change in Optical Coherence Tomography (OCT) central subfield retinal thickness (CST) from baseline by visit over time
Time Frame: Day 1 to Week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
Microns
  Week 8: number analyzed (Participants) | 127 | 123
  Week 8 | -9.8 (10.64) | 4.5 (17.22)
  Week 20: number analyzed (Participants) | 122 | 109
  Week 20 | -12.8 (13.42) | 6.6 (28.99)
  Week 32: number analyzed (Participants) | 117 | 99
  Week 32 | -13.9 (14.88) | 5.2 (27.86)
  Week 44: number analyzed (Participants) | 109 | 90
  Week 44 | -8.9 (19.71) | -0.5 (17.12)
  Week 48: number analyzed (Participants) | 114 | 91
  Week 48 | -15.2 (16.35) | -0.7 (15.76)

15. Other Pre Specified Outcome: Mean Change in BCVA
Description: Mean change in Best-corrected Visual Acuity (BCVA) from baseline by visit over time. Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA letter score from baseline indicates an improvement in visual acuity.
Time Frame: Day 1 to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | KSI-301 - Treatment Group A | Treatment Group B
Number analyzed (Participants) | 128 | 125
ETDRS Letters
  Week 8: number analyzed (Participants) | 127 | 123
  Week 8 | 1.3 (5.02) | 0.2 (4.80)
  Week 20: number analyzed (Participants) | 122 | 109
  Week 20 | 1.1 (5.22) | 0.3 (6.29)
  Week 32: number analyzed (Participants) | 117 | 99
  Week 32 | 0.9 (8.68) | 1.2 (4.87)
  Week 44: number analyzed (Participants) | 109 | 90
  Week 44 | 1.0 (5.63) | 1.6 (5.55)
  Week 48: number analyzed (Participants) | 114 | 91
  Week 48 | 1.1 (6.44) | 1.5 (5.49)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported through the End of Study or Early Termination (ET)
Description: The "At Risk" numbers for "post Week 48 to the end of study" columns are number of participants who continued in the study after Week 48 from the Participant Flow.
Groups:
- KSI-301 - Treatment Group A (Day 1 to Week 48); KSI-301 - Treatment Group A (Post Week 48 to End of Study): Intravitreal injection of KSI-301 (5 mg): three initiating doses, and then every 24 weeks through Week 92
  KSI-301: Intravitreal injection
- Treatment Group B (Day 1 to Week 48); Treatment Group B (Post Week 48 to End of Study): Sham injection on the same schedule as Treatment Group A
  Sham injection: The sham injection is a procedure that mimics an intravitreal injection. It involves pressing the blunt end of an empty syringe (without a needle) against the anesthetized eye. It is performed to maintain masking of the study.
Arm/Group | KSI-301 - Treatment Group A (Day 1 to Week 48) | Treatment Group B (Day 1 to Week 48) | KSI-301 - Treatment Group A (Post Week 48 to End of Study) | Treatment Group B (Post Week 48 to End of Study)
All-Cause Mortality (participants affected / at risk) | 1/128 | 1/125 | 1/120 | 0/115
Serious Adverse Events (participants affected / at risk) | 18/128 | 12/125 | 8/120 | 3/115
Other Adverse Events (participants affected / at risk) | 49/128 | 51/125 | 15/120 | 9/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 - Treatment Group A (Day 1 to Week 48) (N=128) | Treatment Group B (Day 1 to Week 48) (N=125) | KSI-301 - Treatment Group A (Post Week 48 to End of Study) (N=120) | Treatment Group B (Post Week 48 to End of Study) (N=115)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion - Fellow Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSI-301 - Treatment Group A (Day 1 to Week 48) (N=128) | Treatment Group B (Day 1 to Week 48) (N=125) | KSI-301 - Treatment Group A (Post Week 48 to End of Study) (N=120) | Treatment Group B (Post Week 48 to End of Study) (N=115)
Cataract - Study Eye (Eye disorders) | 13 (14) | 5 (5) | 3 (3) | 0 (0)
Conjunctival haemorrhage - Study Eye (Eye disorders) | 9 (9) | 4 (5) | 1 (1) | 0 (0)
Cataract - Fellow Eye (Eye disorders) | 7 (7) | 3 (3) | 1 (1) | 0 (0)
Diabetic retinal oedema - Study Eye (Eye disorders) | 2 (2) | 18 (19) | 3 (3) | 3 (3)
Diabetic retinopathy - Study Eye (Eye disorders) | 2 (2) | 8 (8) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 9 (9) | 6 (7) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 15 (15) | 8 (8) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 12 (13) | 10 (10) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT05066230/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT05066230/SAP_001.pdf